CLINICAL TRIAL: NCT02320604
Title: Pharmacokinetics of Liposomal Amphotericin B (AmBisome®) Given Intravenously to Patients Undergoing Bariatric Surgery
Brief Title: Liposomal Amphotericin B (AmBisome) Pharmacokinetics Given as a Single Intravenous Dose to Obese Patients (ASPEN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UMCN-AKF 14.04
Record Dates: First submitted 2014-10-31; First posted 2014-12-19 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2019-01

CONDITIONS: Morbid Obesity
Keywords: Liposomal amphotericin B; AmBisome; Pharmacokinetics; Obesity; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese Subjects 1mg/kg (Experimental): 8 obese subjects will receive 1mg/kg Ambisome i.v. infused over 45 minutes
  Interventions: Drug: Administration of study drug
- Obese Subjects 2mg/kg (Experimental): 8 obese subjects will receive 2mg/kg Ambisome i.v. infused over 90 minutes
  Interventions: Drug: Administration of study drug

INTERVENTIONS:
Drug: Administration of study drug — i.v. administration of Ambisome in two different dossages
  Other Names: Ambisome

SUMMARY:
Dosing guidelines for liposomal amphotericin B (AmBisome) in (morbidly) obese patients are not available. Subsequently, the pharmacokinetic profile of AmBisome in this specific patient population is still largely unknown.

To build a valid pharmacokinetic model, obese patients with a BMI ≥ 40 undergoing endoscopic gastric bypass surgery will receive a single dose of 1 mg/kg or 2 mg/kg AmBisome (besides standard anti-bacterial prophylaxis) and a PK-curve will be drawn. These PK-values can then be compared to the pharmacokinetics of a normal-weight group.

DETAILED DESCRIPTION:
* The overall trial design is a prospective, open-label, non-randomized, single-centre, single-dose, multiple dose level trial, (1 mg/kg and 2 mg/kg).
* A total of sixteen patients with a BMI ≥40 kg/m2 undergoing bariatric surgery who receive a pre-surgery dose of AmBisome 1 mg/kg (n=8) or 2 mg/kg (n=8) will be enrolled.
* After enrollment of group 1 (1 mg/kg), an interim analysis on the safety of AmBisome will be performed before proceeding to group 2 (2 mg/kg).
* Infusion time and concentration of AmBisome will be 45 minutes (1 mg/kg group) and 90 minutes (2 mg/kg group)
* A PK curve will be determined after administration of a single, pre-surgery dose of AmBisome at t = 0.5, 0.75 (end of infusion group 1), 1.5 (end of infusion group 2), 2, 4, 6, 8, 10, 12, 24, 36, and 48 and (if feasible) 72 hours post infusion (n=12 samples) for group 1 (1 mg/kg), 8 patients.The PK curve of group 2 (2 mg/kg, 8 patients) will be similar to group 1, except for the t=1.5 hour sampling point, which will be end of infusion due to the infusion time of 90 minutes.
* Patients are considered to have completed the study if at least 9/11 samples of the PK curve up until 48 hours have been collected.
* Patients will be selected by the research team to have a good spread in weight bands.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a BMI ≥40 kg/m2 and is undergoing bariatric surgery
2. Subject is at least 18 of age on the day of screening.
3. Subject or legal representatives are able and willing to sign the Informed Consent before screening evaluations.

Exclusion Criteria:

1. Documented history of sensitivity to medicinal products or excipients similar to those found in the polyene preparation.
2. History of, or current abuse of drugs, alcohol or solvents (up until a maximum of three months before enrolment).
3. Inability to understand the nature of the trial and the procedures required.
4. Administration of nephrotoxic medication (aminoglycosids, immunosuppressants, antivirals, antineoplastic agents) up until a maximum of one month before enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) 0-inf Ambisome | at t = 0.5, 0.75, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 and (if feasible) 72 hours post infusion
  The primary outcome measurement will be the area under the plasma concentration-time curve (AUC) from time 0 to infinitive (inf) post infusion (AUC0- inf) value of AmBisome. This will be determined by use of the log-linear trapezoidal rule.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) Ambisome | at t = 0.5, 0.75, 1.5, 2, 4, 6, 8, 10, 12, 24, 36 and 48 and (if feasible) 72 hours post infusion
  Peak concentration over the sampling interval.

CONTACTS AND LOCATIONS:
Overall Officials: Roeland E Wasmann, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - St. Antonius hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No
No plan has been made. Individual researchers are welcome to request data with our group.

REFERENCES:
- [Background] Wasmann RE, Smit C, van Dongen EPH, Wiezer RMJ, Adler-Moore J, de Beer YM, Burger DM, Knibbe CAJ, Bruggemann RJM. Fixed Dosing of Liposomal Amphotericin B in Morbidly Obese Individuals. Clin Infect Dis. 2020 May 6;70(10):2213-2215. doi: 10.1093/cid/ciz885. PMID 31588493
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/31588493/